CLINICAL TRIAL: NCT04300595
Title: The Efficacy of Combined Local and General Anesthesia or General Anesthesia Alone in External Dacryocystorhinostomy: A Randomized Controlled Study
Brief Title: Anesthetic Approaches for Dacryocystorhinostomy Surgery: The Effect of Adding Local Anesthesia to General Inhalational Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Mohamed EL -Asser,MD, Heba Mohamed EL -Asser,MD, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: local anesthesia in DCR
Record Dates: First submitted 2020-02-17; First posted 2020-03-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Effects of; Anesthesia, Local,Pain,in DISE
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: The day before surgery and after obtaining written informed consent and full history taking, all patients were assigned randomly to receive either general anesthesia with intravenous opioids and local infiltration of saline (Group G) or general anesthesia with intravenous saline and local infiltration of a mixture of lidocaine/epinephrine (Group L).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the Group G, Local infiltration of 10 ml normal saline at site of skin incision after marking and analgesia was provided by 40 µg/kg nalbuphine loaded in 10 ml syringe IV before skin incision and subsequent injections of 10-20 µg/kg nalbuphine as necessary. The last supplemental bolus of nalbuphine was given at least 30 min before the end of the operation In the Group L, Local infiltration of 10 ml mixture of 20 mg/ml lidocaine and 10 µg/ml epinephrine (instead of saline used in Group G) and normal saline in 10 ml syringe was given IV (instead of nalbuphine used in Group G).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia (Group G) (Active Comparator): Patients receive general anesthesia with intravenous opioids and local infiltration of saline (Group G)
  Interventions: Procedure: Combination of General anesthesia and local anesthesia in dacryocystorhinostomy surgery
- Local anesthesia (Group L) (Active Comparator): Patients receive general anesthesia with intravenous saline and local infiltration of a mixture of lidocaine/epinephrine (Group L).
  Interventions: Procedure: Combination of General anesthesia and local anesthesia in dacryocystorhinostomy surgery

INTERVENTIONS:
Procedure: Combination of General anesthesia and local anesthesia in dacryocystorhinostomy surgery — all patients were assigned randomly to receive either general anesthesia with intravenous opioids and local infiltration of saline (Group G) or general anesthesia with intravenous saline and local infiltration of a mixture of lidocaine/epinephrine (Group L).
  In both groups, general anesthesia was induced with 2 mg/kg propofol and tracheal intubation was facilitated by 0.1 mg/kg cisatracurium. All patients underwent mechanical ventilation with 100% oxygen. Anesthesia was maintained with isoflurane, and muscle relaxation was provided by an injection of cisatracurium 0.02 mg/kg every 20 minutes.

SUMMARY:
To Study the effect of combination of of general anesthesia and local anesthesia in anesthesia for external dacryocystorhinostomy and assess quality of the procedure

DETAILED DESCRIPTION:
* calculate the total requirement for anaesthetic agents to maintain satisfactory operating conditions
* calculate total anesthetic time
* assess intraoperative changes in hemodynamics
* assess intraoperative blood loss
* evaluate surgeon and patient satisfaction
* recognize whether this was related with changes in postoperative analgesia .
* Also occurrence of postoperative nausea was recorded and compared with general anaesthesia combined with intravenous opioid for (EXT-DCR) surgery.

ELIGIBILITY:
Inclusion Criteria:• Age from 20 to 50 years old.

* American society of anesthesiologists (ASA) physical status I or II.
* Elective unilateral Dacryocystorhinostomy with paranasal skin incision.

Exclusion Criteria:

* Endoscopic Dacryocystorhinostomy.
* Allergy to amide local anesthetics or opioids.
* Drug abuse.
* Pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain assessment | change in visual analogue scale at 1, 2, 4, 6, 8, 12, and 24 hours postoperative after extubation
  To quantify the intensity of postoperative pain, the patients were asked to use a 10-cm visual analog scale (VAS) grade from 0-cm (no pain) to 10-cm (the worst possible pain) 1, 2, 4, 6, 8, 12, and 24 h after extubation
hemodynamic assessment | for 24 hours
  Change in heart rate were recorded preoperatively, after induction of general anesthesia, after IV injection of 10 ml syringe and after local infiltration, then every 5 min intraoperatively, and during early recovery, and every 30 min, thereafter for 24 hours
hemodynamic assessment | for 24 hours
  Change in arterial blood pressure were recorded preoperatively, after induction of general anesthesia, after IV injection of 10 ml syringe and after local infiltration, then every 5 min intraoperatively, and during early recovery, and every 30 min, thereafter for 24 hours

SECONDARY OUTCOMES:
extubation time | intraoperative (from time of anesthesia ended till extubation and recorded in each patient in minutes)
  Extubation time was calculated from time of anesthesia off till extubation and recorded in each patient
mean isoflurane % | intraoperative ( recorded every 5 minutes)
  Isoflurane concentration was adjusted according to hemodynamics by increase or decrease concentration when heart rate or mean arterial blood pressure increase or decrease more than 20-30% of the basal preoperative record, respectively and after nalbuphine dose failed to adjust hemodynamics
time to rescue analgesia | up to 24 hours of postoperative
  The time from the end of anaesthesia to ﬁrst use of rescue analgesia (nalbuphine)
The number of patients who required nalbuphine in the postoperative period, | up to 24 hours of postoperative
  to calculate the number of patients who required nalbuphine in the postoperative period,
intraoperative bleeding | at the end of surgery
  to the nearest milliliter) was determined by the amount of blood in the suction containers and gauze sponges, based on assessment by the surgeon.
patient and surgeon satisfaction | assessed on the first postoperative day from both patients and surgeons.
  An overall satisfaction score according to postoperative analgesia .
  * nil = 0
  * mild = 1
  * good = 2
  * excellent = 3 was recorded on the first postoperative day from both patients and surgeons. The acceptance of combination of LA and GA was questioned and the patients who applied for a successive operation on the other eye were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Heba M EL-Asser, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scawn RL, Allen MJ, Rose GE, Verity DH. Randomised, masked study of local anaesthesia administered prior to external dacryocystorhinostomy under general anaesthesia. Eye (Lond). 2019 Mar;33(3):374-379. doi: 10.1038/s41433-018-0201-5. Epub 2018 Sep 18. PMID 30228368
- [Background] Ghali AM, El Btarny AM. The effect on outcome of peribulbar anaesthesia in conjunction with general anesthesia for vitreoretinal surgery. Anaesthesia. 2010 Mar;65(3):249-53. doi: 10.1111/j.1365-2044.2009.06191.x. Epub 2009 Dec 23. PMID 20039868